CLINICAL TRIAL: NCT01135134
Title: Multicenter, Double-blind, Randomized, Placebo-controlled Study of Mometasone Furoate Nasal Spray in Pediatric Subjects With Perennial Allergic Rhinitis (Protocol No.P06332)
Brief Title: Multicenter, Double-blind, Randomized, Placebo-controlled Study of Mometasone Furoate Nasal Spray in Pediatric Subjects With Perennial Allergic Rhinitis (Study P06332)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P06332
Record Dates: First submitted 2010-05-28; First posted 2010-06-02 (Estimated); Results first posted 2011-11-03 (Estimated); Last update posted 2024-05-28 (Actual); Status verified 2022-02

CONDITIONS: Rhinitis, Allergic, Perennial
MeSH Terms: conditions — Rhinitis, Allergic, Perennial | interventions — Mometasone Furoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mometasone furoate nasal spray (MFNS) (50 μg spray device) (Experimental): The dose will be as follows:
  * 5 to 11 years: one spray per nostril once daily (100 μg/day as MF) in the morning for 2 weeks
  * 12 to 15 years: 2 sprays per nostril once daily (200 μg/day as MF) in the morning for 2 weeks
  Interventions: Drug: Mometasone furoate
- MF placebo nasal spray (Placebo Comparator): Administration will be as follows:
  * 5 to 11 years: one spray per nostril once daily in the morning for 2 weeks
  * 12 to 15 years: 2 sprays per nostril once daily in the morning for 2 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mometasone furoate — The study drug is MFNS (50 μg spray device) and the dose will be:
  * 5 to 11 years: one spray per nostril once daily (100 μg/day as MF) in the morning for 2 weeks
  * 12 to 15 years: 2 sprays per nostril once daily (200 μg/day as MF) in the morning for 2 weeks
  Other Names: Nasonex
  Arms: Mometasone furoate nasal spray (MFNS) (50 μg spray device)
Drug: Placebo — MF Placebo nasal spray and administration will be as follows:
  * 5 to 11 years: one spray per nostril once daily in the morning for 2 weeks
  * 12 to 15 years: 2 sprays per nostril once daily in the morning for 2 weeks
  Arms: MF placebo nasal spray

SUMMARY:
This is a multicenter, randomized, parallel design, double-blind study of mometasone furoate (MF) in pediatric subjects with perennial allergic rhinitis. The subjects 5 to 15 years of age with perennial allergic rhinitis will enter a no-treatment observation period of 7 days at minimum and eligibility for inclusion in this study will be assessed. Following the observation period, eligible subjects will be randomized to MF or MF placebo for a 2-week double-blind treatment. At each clinic visit (at the start of treatment and after 1 and 2 weeks of treatment or at discontinuation), nasal symptom scores, nasal findings, and adverse events (AEs), will be evaluated. A 30-day follow-up visit will take place after the completion (or discontinuation) of the 2-week treatment period, to confirm presence or absence of serious adverse events (SAEs) and trial procedure-related AEs.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric subjects with perennial allergic rhinitis who satisfy all of the following main criteria:

  * Subjects having symptoms of perennial allergic rhinitis of moderate to severe degree, after the pretreatment observation period.
  * Subjects confirmed to be allergic to non-seasonal environmental antigens (e.g., house dust-mite antigen).
  * Male or female outpatients aged 5 to 15 years at the time of providing informed consent.

Exclusion Criteria:

* Subjects for whom any of the main exclusion criteria below is applicable will not be registered in this study.

  * Subjects with coexisting tuberculous disease or lower respiratory tract infection and subjects who have a nasopharyngolaryngeal infection (acute upper respiratory tract infection, acute pharyngolaryngitis, or acute tonsillitis, etc.) requiring treatment at the time of registration
  * Subjects with coexisting infections or systemic mycosis for which there are no effective antibiotics
  * Subjects with repeated epistaxis
  * Subjects who have nasal septum ulcers, nasal surgery, or nasal trauma, which have not healed
  * Subjects with severe hepatic, renal, cardiac, hematological disease, diabetes mellitus, hypertension, or other serious coexisting diseases and whose general condition is poor
  * Subjects with complication of vasomotor rhinitis or eosinophilic rhinitis.
  * Subjects with nasal conditions (infectious sinusitis, hypertrophic rhinitis, acute or chronic rhinitis, nasal polyps, septal deviation, etc.) which may interfere with the evaluation of the efficacy of the study drug.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 333 (Actual)
Dates: Start 2010-06; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Okamoto Y, Suzuki I . Multicenter, double-blind, randomized, placebo-controlled study of mometasone furoate nasal spray in Japanese pediatric subjects with perennial allergic rhinitis . Oto-rhino Laryngol Tokyo. 2013;106(11):1045-1057.

RESULTS

PARTICIPANT FLOW:
Groups:
- MFNS: Mometasone furoate nasal spray (MFNS) 50 mcg nasal spray device. The dose was as follows:
  * 5 to 11 years: one spray per nostril once daily (100 mcg/day as MF) in the morning for 2 weeks.
  * 12 to 15 years: 2 sprays per nostril once daily (200 mcg/day as MF) in the morning for 2 weeks.
- Placebo: Placebo MFNS. Administration was as follows:
  * 5 to 11 years: one spray per nostril once daily in the morning for 2 weeks.
  * 12 to 15 years: 2 sprays per nostril once daily in the morning for 2 weeks.
Period: Overall Study
Arm/Group | MFNS | Placebo
Started | 220 | 113
Completed | 218 | 112
Not Completed | 2 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Did not meet protocol eligibility | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MFNS | Placebo | Total
Number analyzed (Participants) | 220 | 113 | 333
Age, Customized [Number; unit: Participants]
  Between 5 and 11 years | 146 | 74 | 220
  Between 12 and 15 years | 74 | 39 | 113
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 38 | 128
  Male | 130 | 75 | 205

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Total Nasal Symptom Score at 2 Weeks
Description: Total nasal symptom score was a composite of 4 symptoms (sneezing, rhinorrhea, nasal congestion, and nasal itching), each symptom was scored on a scale of 0 = none, 1 = mild, 2 = moderate, 3 = severe. The total score ranged from 0 to 12. The higher the score was, the more severe the symptoms were.
Time Frame: Baseline and 2 weeks (or discontinuation)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | MFNS | Placebo
Number analyzed (Participants) | 220 | 113
score on a scale | -3.9850 (0.1633) | -1.9081 (0.2233)
Statistical Analysis 1: Comparison: MFNS vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA

2. Secondary Outcome: Change From Baseline in the Total Nasal Symptom Score at 1 Week
Description: as for outcome 1
Time Frame: Baseline and 1 week
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | MFNS | Placebo
Number analyzed (Participants) | 219 | 113
score on a scale | -2.4686 (0.1441) | -1.1651 (0.1967)
Statistical Analysis 1: Comparison: MFNS vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA

ADVERSE EVENTS:
Arm/Group | MFNS | Placebo
Serious Adverse Events (participants affected / at risk) | 0/220 | 0/113
Other Adverse Events (participants affected / at risk) | 24/220 | 19/113
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MFNS (N=220) | Placebo (N=113)
Naspharyngitis (Infections and infestations) | 11 (11) | 10 (10)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 13 (15) | 11 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to provide to the Sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the trial. The Sponsor shall have the right to review and comment with respect to publications, abstracts, slides, and manuscripts and the right to review and comment on the data analysis and presentation.